CLINICAL TRIAL: NCT04540159
Title: Measurement of Immune Checkpoints in Intraabdominal Ascites Fluid in Patients With Advanced Colorectal Cancer
Brief Title: Immune Checkpoints in Intraabdominal Ascites Fluid
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Other Study IDs: Colorectal Checkpoints
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: Ascites; Immune checkpoints; Flow-cytometry
MeSH Terms: conditions — Colorectal Neoplasms; Ascites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Advanced stage Colorectal cancer patients with intraabdominal ascites
  Interventions: Diagnostic Test: Flow-cytometric analysis
- Control: Liver cirrhosis and congestive heart failure patients with intraabdominal ascites
  Interventions: Diagnostic Test: Flow-cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow-cytometric analysis — Measuring the level of sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9 in the intraabdominal ascites

SUMMARY:
Colorectal cancers are the third most common type of cancer in the world. Peritoneal carcinomatosis and intraabdominal acid development occur in advanced stages of colorectal cancers.

It is known that the immune system plays an important role in tumor development or tumor eradication. Among the mechanisms of escape from the immune system, changes in the tumor microenvironment play an important role.

Immune checkpoints are molecules that have become popular especially after the Nobel Prize in 2018, and are important in revealing the relationship between cancer and the immune system.

In our study, it is aimed to evaluate whether there is a difference in intraabdominal ascites fluid immune checkpoints level in patients with advanced colorectal cancer patients compared to patients without malignancy.

DETAILED DESCRIPTION:
Colorectal cancers are the third most common type of cancer in the world. Peritoneal carcinomatosis and intraabdominal acid development occur in advanced stages of colorectal cancers.

It is known that the immune system plays an important role in tumor development or tumor eradication. The role of the immune system in colorectal cancers has been demonstrated with the effects of tumor-infiltrating lymphocytes (TIL) and immune control points on TILs or immune control point ligands on patient survival, especially in recent studies. Studies in the literature usually include immunological examinations of patient blood or tumor tissue.

Immune checkpoints are molecules that have become popular especially after the Nobel Prize in 2018, and are important in revealing the relationship between cancer and the immune system. Programmed Cell Death Protein-1 (PD-1) and its ligand, PD-L1, is an immune checkpoint that acts by blocking T cell receptor signal transduction and auxiliary stimuli. T cell immunoglobulin and mucin domain 3 (TIM-3) are mostly expressed on T cells, Tregs, dendritic cells, B cells, macrophages, natural killer cells (NK) and mast cells that produce interferon-(10). Impairment in regulation of TIM-3 expression has been associated with autoimmune diseases. High TIM-3 expression is associated with suppression of T cell responses and T cell depletion, which is characterized by loss of T cell functions during chronic viral infections and during tumor development. With the clinical success of immune checkpoint inhibitors such as ipilimumab and nivolumab for melanoma and lung cancer, immune checkpoints have attracted more attention.

There are many publications in the literature evaluating immunological markers from ascites fluid samples for various reasons. In these studies, T and B cell subtypes were examined from ascites fluid samples taken from patients with ascites, especially ovarian cancer and liver cirrhosis. In the only study on gastrointestinal cancers, immunophenotyping was performed in intraabdominal ascites and blood in 22 advanced gastrointestinal tumor patients and some cell subgroups were associated with worse clinical outcome. In the literature, there is no study on cytokine analysis from intra-abdominal ascites fluids specific to colorectal cancer.

In our study, it is aimed to evaluate whether there is a difference in intraabdominal ascites fluid immune checkpoints level in patients with advanced colorectal cancer patients compared to patients without malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage colorectal cancer patients with intraabdominal ascites

Exclusion Criteria:

* Patients who have cancer other than colorectal cancer
* Patients with peritonitis
* Pregnant women
* HIV (+) patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ergegadfgegrr
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Immune Checkpoint levels | 4 months
  Measuring the level of sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9 in the intraabdominal ascites

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Ufuk Oguz Idiz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakano M, Ito M, Tanaka R, Yamaguchi K, Ariyama H, Mitsugi K, Yoshihiro T, Ohmura H, Tsuruta N, Hanamura F, Sagara K, Okumura Y, Nio K, Tsuchihashi K, Arita S, Kusaba H, Akashi K, Baba E. PD-1+ TIM-3+ T cells in malignant ascites predict prognosis of gastrointestinal cancer. Cancer Sci. 2018 Sep;109(9):2986-2992. doi: 10.1111/cas.13723. PMID 30187676
- [Background] Radestad E, Klynning C, Stikvoort A, Mogensen O, Nava S, Magalhaes I, Uhlin M. Immune profiling and identification of prognostic immune-related risk factors in human ovarian cancer. Oncoimmunology. 2018 Nov 16;8(2):e1535730. doi: 10.1080/2162402X.2018.1535730. eCollection 2019. PMID 30713791
- [Background] Yoshida N, Kinugasa T, Miyoshi H, Sato K, Yuge K, Ohchi T, Fujino S, Shiraiwa S, Katagiri M, Akagi Y, Ohshima K. A High RORgammaT/CD3 Ratio is a Strong Prognostic Factor for Postoperative Survival in Advanced Colorectal Cancer: Analysis of Helper T Cell Lymphocytes (Th1, Th2, Th17 and Regulatory T Cells). Ann Surg Oncol. 2016 Mar;23(3):919-27. doi: 10.1245/s10434-015-4923-3. Epub 2015 Nov 12. PMID 26564244